CLINICAL TRIAL: NCT03212716
Title: Validation of the Efficiency of Molecules Reproposed on the Basis of Their Cellular Transcriptomic Signature, Antagonist of the Signature Determined in Infection Due to Virus Influenza A.
Brief Title: Efficiency of Antagonist Drugs of the Cellular Transcriptomic Signature of Influenza A Virus Infection.
Acronym: FLUNEXT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: rate of inclusion and study affected by covid-19 epidemic
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015_65; 2016-004222-42 (EudraCT Number); PHRC_N -15-0442 (Other: PHRC number)
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Flu
Keywords: Infectiology; Biology of infectious agents; Flu; Intensive care
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Diltiazem

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diltiazem (Experimental): oseltamivir + diltiazem
  Interventions: Drug: Oseltamivir; Drug: Diltiazem
- oseltamivir + placebo (Placebo Comparator): oseltamivir + placebo of diltiazem
  Interventions: Drug: Oseltamivir; Drug: Placebos

INTERVENTIONS:
Drug: Oseltamivir — 150 mg twice a day during 10 days (ANSM guidelines for severe flu).
Drug: Diltiazem — 60 mgx3 per day during 10 days.
  Arms: diltiazem
Drug: Placebos — Placebo of diltiazem
  Arms: oseltamivir + placebo

SUMMARY:
The aim of this study is to evaluate the possibility to repropose marketed drugs as antiviral ones, based on their ability to reverse the transcriptomic signature of the infected cells. This strategy has to be considered is the context of emerging viral diseases and of increase of resistance to antivirals. Concerning infection by Influenza viruses, the main drugs were identified and evaluated on in vitro and in vivo models: diltiazem. Therefore, it will be assess the efficacy of these the drug, compared to placebo, to treat severe flu.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in intensive care units,
* patients with mechanical ventilation invasive or non-invasive or Optiflow® ventilation system.
* for a suspicion of severe flu,
* with a symptoms for less than 96 hours,
* and a respiratory failure defined by the necessity to resort to mechanical ventilation, invasive or Optiflow® Ventilation System The inclusion is conditioned to the detection of Influenza A viruses by PCR on nasopharyngeal swab.

Exclusion Criteria:

* No consent.
* Hypersensibility to Oseltamivir
* Negative PCR on nasopharyngeal swab
* Symptoms for more than 96 hours.
* Moribund patients at inclusion.
* Pregnant/nursing woman.
* Patients already taking diltiazem in the 48 hours before.
* Patients having taken more than 3 intakes of oseltamivir before randomization.
* Hemodynamic instability needing a dose of noradrenaline exceeding 2mg/h

Contraindication to diltiazem:

* sinusal dysfunction without device.
* auriculo-ventricular heart block without device.
* Cardiogenic pulmonary oedema.
* Left cardiac failure
* bradycardia<40/min
* Concomitant use of beta-blockers, antiarrythmic drugs, especially amiodarone.
* Concomitant use of ivabradine, pimozide, nifedipine, ergot alkaloids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Percentage of alive patients without detection of influenza A virus by RT-PCR in nasopharyngeal swabs, | 7 days after the beginning of the treatment.

SECONDARY OUTCOMES:
Delay needed for the negativation of influenza A detection by RT-PCR | up to 10days
Overall mortality | At 28 days
Length of mechanical ventilation | an average of 10 days
Change in Oxygenation (PaO2/FiO2 Ratio) | once day for 10 days and at 28 days
  Arterial blood samples for blood gas analysis are collected during the treatment period. The differences in the mean values of PaO2/FiO2 ratio are registered and analysed.
Length of hospitalization | an average of 10 days in ICU and of 16 days in hospital
Length of extracorporeal membrane oxygenation (ECMO) if implemented. | an average of 10 days
Transcriptomic signature determined by the DNA microarray technology and analysed by bioinformatic tools | Four time points : at inclusion, the first day after inclusion, the fourth day after inclusion, and the seventh day after inclusion
  evaluation of the capacity of tested molecules to reverse the transcriptomic signature linked to the viral infection

CONTACTS AND LOCATIONS:
Overall Officials: Julien Poissy, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (19):
- France (19):
  - Chu Amiens Picardie, Amiens
  - CH ARRAS, Arras
  - Ch Hnfc Site de Belfort, Belfort
  - Ch Bethune, Béthune
  - Ch Pierre Oudot Bourgoin Jallieu, Bourgoin
  - Chru Brest, Brest
  - CH DOUAI, Douai
  - Hôpital Raymond Poincaré, Garches
  - CH LENS, Lens
  - Hôpital Roger Salengro, CHRU, Lille
  - Hôpital Edouard Herriot Hospices Civils de Lyon, Lyon
  - CH de Montauban, Montauban
  - Ch Regional Orleans, Orléans
  - Gpe Hosp Cochin Saint Vincent de Paul - Paris, Paris
  - Hu Paris Sud Site Kremlin Bicetre Aphp, Paris
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Bretonneau, Tours
  - Ch de Valenciennes, Valenciennes
  - Centre Hospitalier de Versailles - Le Chesnay Rocquencourt, Versailles